CLINICAL TRIAL: NCT05170321
Title: Analysis of Influencing Factors and Construction of Prediction Models of Artificial Joint Replacement in China
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: 2017121016
Record Dates: First submitted 2021-12-08; First posted 2021-12-27 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-11

CONDITIONS: Knee Arthropathy; Hip Arthropathy; Shoulder Arthropathy; Ankle Arthropathy; Elbow Arthropathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- patients undergoing knee arthroplasty in Hospital Quality Monitoring System in China: Patients who underwent knee arthroplasty and was recorded in HQMS were included in this group
- patients undergoing hip arthroplasty in Hospital Quality Monitoring System in China: Patients who underwent hip arthroplasty and was recorded in HQMS were included in this group
- patients undergoing shoulder arthroplasty in Hospital Quality Monitoring System in China: Patients who underwent shoulder arthroplasty and was recorded in HQMS were included in this group
- patients undergoing ankle arthroplasty in Hospital Quality Monitoring System in China: Patients who underwent ankle arthroplasty and was recorded in HQMS were included in this group
- patients undergoing elbow arthroplasty in Hospital Quality Monitoring System in China: Patients who underwent elbow arthroplasty and was recorded in HQMS were included in this group

SUMMARY:
The project intends to analyze the epidemiological characteristics, risk factors, complications and resource utilization of artificial joint replacement in China through the inpatient data collected by the Hospital Quality Monitoring System (HQMS). The HQMS database is a mandatory electronic inpatient database system developed by the National Health Commission of the People's Republic of China. Since 2013, tertiary hospitals have been required to upload their inpatient discharge records. By 2019, the HQMS database has included more than 230 million standardized inpatient discharge records of over 1000 hospitals across all 31 provincial-level administrative regions in mainland China. Patient demographics, clinical diagnosis, procedures and operations, drug use, costs and complications were all recorded in the HQMS database. The investigators planned to include five types of arthroplasty, including knee arthroplasty, hip arthroplasty, shoulder arthroplasty, ankle arthroplasty and elbow arthroplasty. The data analysis will be conformed to the principle of confidentiality and will not reveal the privacy of those patients. The data will be only used for this research project and there is no conflict of interest. It is in line with the principles of ethics, harmlessness and fairness. This study was authorized by the HQMS Committee Board and approved by the institutional review board, with waiver of informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent knee, hip, shoulder, ankle and elbow arthroplasty in HQMS

Exclusion Criteria:

* Patients who didn't undergo knee, hip, shoulder, ankle and elbow arthroplasty
* Patients with missing demographics or medical data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent knee, hip, shoulder, ankle and elbow arthroplasty were included.
Sampling Method: Non-Probability Sample
Enrollment: 600000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Epidemiological characteristics, complications, risk factors and resource utilization of knee arthroplasty in China | 10 years (2013-2022)
  The project intends to analyze the epidemiological characteristics, complications, risk factors and resource utilization of artificial knee joint replacement in China through the inpatient data collected by the Hospital Quality Monitoring System (HQMS). The information collected by HQMS includes demographics characteristics, hospitalization information, medical care cost, complications, et al.
Epidemiological characteristics, complications, risk factors and resource utilization of hip arthroplasty in China | 10 years (2013-2022)
  The project intends to analyze the epidemiological characteristics, complications, risk factors and resource utilization of artificial hip joint replacement in China through the inpatient data collected by the Hospital Quality Monitoring System (HQMS). The information collected by HQMS includes demographics characteristics, hospitalization information, medical care cost, complications, et al.
Epidemiological characteristics, complications, risk factors and resource utilization of shoulder arthroplasty in China | 10 years (2013-2022)
  The project intends to analyze the epidemiological characteristics, complications, risk factors and resource utilization of artificial shoulder joint replacement in China through the inpatient data collected by the Hospital Quality Monitoring System (HQMS). The information collected by HQMS includes demographics characteristics, hospitalization information, medical care cost, complications, et al.
Epidemiological characteristics, complications, risk factors and resource utilization of ankle arthroplasty in China | 10 years (2013-2022)
  The project intends to analyze the epidemiological characteristics, complications, risk factors and resource utilization of artificial ankle joint replacement in China through the inpatient data collected by the Hospital Quality Monitoring System (HQMS). The information collected by HQMS includes demographics characteristics, hospitalization information, medical care cost, complications, et al.
Epidemiological characteristics, complications, risk factors and resource utilization of elbow arthroplasty in China | 10 years (2013-2022)
  The project intends to analyze the epidemiological characteristics, complications, risk factors and resource utilization of artificial elbow joint replacement in China through the inpatient data collected by the Hospital Quality Monitoring System (HQMS). The information collected by HQMS includes demographics characteristics, hospitalization information, medical care cost, complications, et al.

CONTACTS AND LOCATIONS:
Overall Officials: Guanghua Lei, PhD; MD, Principal Investigator — Xiangya Hospital
Locations (1):
- Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No
The investigators do not wish to share our data according to the policy of our hospital, the data could not be shared with others without permission.

REFERENCES:
- [Background] Zeng C, Lane NE, Englund M, Xie D, Chen H, Zhang Y, Wang H, Lei G. In-hospital mortality after hip arthroplasty in China: analysis of a large national database. Bone Joint J. 2019 Oct;101-B(10):1209-1217. doi: 10.1302/0301-620X.101B10.BJJ-2018-1608.R1. PMID 31564156
- [Derived] Wang Y, Jiang Q, Long H, Chen H, Wei J, Li X, Wang H, Xie D, Zeng C, Lei G. Trends and benefits of early hip arthroplasty for femoral neck fracture in China: a national cohort study. Int J Surg. 2024 Mar 1;110(3):1347-1355. doi: 10.1097/JS9.0000000000000794. PMID 38320106
- [Derived] Long H, Xie D, Chen H, Wei J, Li X, Wang H, Zeng C, Lei G. Rural-urban differences in characteristics, postoperative outcomes, and costs for patients undergoing knee arthroplasty: a national retrospective propensity score matched cohort study. Int J Surg. 2023 Sep 1;109(9):2696-2703. doi: 10.1097/JS9.0000000000000494. PMID 37247007

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-27): https://cdn.clinicaltrials.gov/large-docs/21/NCT05170321/Prot_SAP_001.pdf